CLINICAL TRIAL: NCT05731245
Title: Efficacy and Safety of Ropeginterferon Alfa-2b for Pre-fibrotic Primary Myelofibrosis and DIPSS Low/Intermediate-1 Risk Myelofibrosis
Brief Title: Ropeginterferon Alfa 2b for Early MyelofibrosisDIPSS Low/Intermediate-1 Risk Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202208080MIPC
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Pre-fibrotic Myelofibrosis
Keywords: Early or Primary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ropeginterferon alfa-2b (Experimental): Eligible subjects will receive ropeg subcutaneously (SC) every 2 weeks at the starting dose of 250µg at week 0, 350 µg at week 2, then 500µg at a fixed dose from week 4 onwards until week 104. In patients achieving a clinical or molecular response at 24 months (week 104), treatment with ropeg will be continued until disease progression.
  Intervention: Drug: Ropeginterferon alfa-2b
  Interventions: Drug: Ropeginterferon Alfa-2B Prefilled Syringe [Besremi]

INTERVENTIONS:
Drug: Ropeginterferon Alfa-2B Prefilled Syringe [Besremi] — Eligible subjects will receive Ropeginterferon alfa-2b subcutaneously (SC) every 2 weeks at the starting dose of 250µg at week 0, 350 µg at week 2, then 500µg at a fixed dose from week 4 onwards

SUMMARY:
This is a multi-centre phase 2 open-label prospective study designed to assess the efficacy and safety of ropeg patients with pre-fibrotic primary myelofibrosis or DIPSS low/intermediate-1 risk myelofibrosis after 24 months of treatment.

DETAILED DESCRIPTION:
This is a multi-centre phase 2 open-label prospective study designed to assess the efficacy and safety of ropeg patients with pre-fibrotic primary myelofibrosis or DIPSS low/intermediate-1 risk myelofibrosis after 24 months of treatment. . In patients achieving any molecular response at 24 months, treatment with ropeg will be continued until disease progression.

After obtaining a written informed consent, screening evaluations will be performed. Eligibility will be determined based on the inclusion and exclusion criteria in section 6 of this protocol. Subject visits will be scheduled regularly after recruitment for efficacy evaluations and safety assessments. A safety follow-up will be scheduled 28 days after end-of-treatment visit. Efficacy evaluations, safety assessments and sample collection will be performed according to the schedule laid in section 2 in this protocol.

Efficacy will be evaluated using laboratory assessment of haematological parameters, physical examination for liver and spleen size assessment, quantitative assessment of JAK2V617F, CALR, MPL and other driver mutations, bone marrow examination, and symptom burden assessment by MPN-SAF-TSS. Quantitative assessment of JAK2V617F, CALR, MPL and other driver mutations will be performed using real-time quantitative PCR or ddPCR at the laboratory at the Department of Medicine, the University of Hong Kong, National Taiwan University Hospital and Chang Gung Memorial Hospital Chiayi.

Safety evaluations will be performed using symptoms, physical examination, laboratory studies, Chest X-rays, ophthalmic assessment, ECOG performance status and CTCAE version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years (or based on the legal age of the territory) Diagnosed of primary myelofibrosis, post-PV and post-ET myelofibrosis according to the WHO 2016 classification Bone marrow reticulin fibrosis grade of 0-1 or low/intermediate-1 risk according to DIPSS Compensated liver function defined as: bilirubin ≤ 1.5 x upper limit normal (ULN); alanine aminotransferase (ALT) ≤ 2 x ULNor aspartate aminotransferase (AST) ≤ 2 x ULN; prothrombin time versus control <3 seconds at screening Glomerular filtration rate ≥ 50 mL/min (by MDRD equation or Cockcroft-Gault formula) Men and women of childbearing potential must agree to perform contraception until 28 days after the last dose of ropeg.

Women must avoid breast-feeding during the study. Able to give a written informed consent and fully comply to the requirements of the study.

Exclusion Criteria:

* Prior or current use of IFNα preparations for PMF or secondary MF. Prior use of IFNα for antecedent PV or ET is allowed provided that the time from the last dose of IFNα to recruitment is > 4 weeks.

Patients currently on other investigational therapy (ies) Contraindications or hypersensitivity to IFNα preparations History of organ transplantation Pregnant or lactating women Documented autoimmune disease at screening Infection with human immunodeficiency virus (HIV) Active and uncontrolled infections with hepatitis B virus (HBV) and hepatitis C virus (HCV). Please note that patients on antiviral therapy with undetectable HBV DNA and HCV RNA may be recruited.

Evidence of severe retinopathy including but not limited to macular degeneration, diabetic retinopathy and hypertensive retinopathy.

History of clinically significant neuropsychiatric conditions including but not limited to depression and epilepsy.

Clinically significant neuropsychiatric conditions including but not limited to depression and epilepsy.

Presence of other active malignancies within three years prior to the time of recruitment. History of malignant disease, including solid tumours and haematological malignancies (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that have been completely excised and are considered cured) within the last 3 years.

Evidence of alcohol or drug abuse within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Clinicohematological responses at 24 weeks | 24 months
  Overall haematological response rate at 6, 12 and 24 months, based on the IWG-MRT and ELN consensus report

SECONDARY OUTCOMES:
Adverse events | 24 months
  Adverse events according to the CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, 100, Taiwan

IPD SHARING:
Plan to Share IPD: No